CLINICAL TRIAL: NCT05405127
Title: Effects of Breathing Exercises With and Without Core Stability Exercises on Pain Pressure Threshold and Disability in Postpartum Females With Lumbopelvic Pain
Brief Title: Breathing and Core Stability Exercise Effects on Lumbopelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0518
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Breathing Sound; Low Back Pain; Post-operative Pain; Pelvic Pain
Keywords: breathing exercises; low back pain; post-partum pain; lumbopelvic pain
MeSH Terms: conditions — Respiratory Sounds; Low Back Pain; Pain, Postoperative; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): breathing exercises
  Interventions: Other: traditional physical therapy
- Core stability exercise (Experimental): core stability exercise along with breathing exercises and pain pressure algometer is used
  Interventions: Other: core stability exercises

INTERVENTIONS:
Other: traditional physical therapy — breathing exercises 10 repetitions, 1set, 3 days/week and targeted abdominal muscles. Total 6 sessions were given each consisting of 30 minutes.
  Arms: Traditional physical therapy
Other: core stability exercises — core stability along with breathing exercise 10 repetitions, 1set, 3 days/week and targeted core muscles. Total 6 sessions were given consisting of 30 minutes.
  Arms: Core stability exercise

SUMMARY:
Lumbopelvic pain refers to self-reported pain in areas of lower region, anterior and posterior pelvic tilt or combination of these. Physical therapy interventions used are breathing exercises with and without core stability exercises. Tool used were Pain Pressure Algometer and Oswestry Disability Index.

DETAILED DESCRIPTION:
Lumbopelvic pain is self-reported pain. It is common complaint for women after labour, and it is found that 25% of newly delivered women experienced low back and pelvic pain. Different interventions have been used to reduce the lumbopelvic pain in general including exercises, drugs, therapies and massage. An increasingly common approach used within physical therapy management are breathing exercises and core stabilization exercises. This study will used to compare the effects of breathing exercises with and without core stability exercise. Pre-assessment will be done using oswestry disability index as subjective measurement and pain pressure algometer as objective measure.

ELIGIBILITY:
Inclusion Criteria:

* Women had parity (2-4) times
* Body mass index that did not exceed 30 Kg/m
* Lumbopelvic pain at least three months until one year postpartum

Exclusion Criteria:

* They were pregnant
* Had systemic inflammatory diseases
* Prolapsed disc
* Neuromuscular disorder

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index | 6th week
  Changes from base line Oswestry disability index was developed first by Fairbank et al. It was designed to measure the back pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100. As the driving section in all the female patients, total score was considered as 45 instead of 50.

SECONDARY OUTCOMES:
Pain Pressure Algometer | 6th week
  Changes from base line Pain Pressure Algometer was developed first by Baba et al. The pressure algometer has linear response to force application between 0 and 1,300 kilopascal.
ROM Back region (flexion) | 6th week
  Changes from the Baseline ROM range of motion of back region flexion was taken.
ROM Back region (extension) | 6th week
  Changes from the baseline ROM range of motion of back region extension was taken.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, MSWHPT, Principal Investigator — Riphah International University
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergstrom C, Persson M, Nergard KA, Mogren I. Prevalence and predictors of persistent pelvic girdle pain 12 years postpartum. BMC Musculoskelet Disord. 2017 Sep 16;18(1):399. doi: 10.1186/s12891-017-1760-5. PMID 28915804
- [Background] Stuber KJ, Wynd S, Weis CA. Adverse events from spinal manipulation in the pregnant and postpartum periods: a critical review of the literature. Chiropr Man Therap. 2012 Mar 28;20:8. doi: 10.1186/2045-709X-20-8. PMID 22455720
- [Background] Gutke A, Lundberg M, Ostgaard HC, Oberg B. Impact of postpartum lumbopelvic pain on disability, pain intensity, health-related quality of life, activity level, kinesiophobia, and depressive symptoms. Eur Spine J. 2011 Mar;20(3):440-8. doi: 10.1007/s00586-010-1487-6. Epub 2010 Jul 1. PMID 20593205
- [Background] Robinson HS, Vollestad NK, Veierod MB. Clinical course of pelvic girdle pain postpartum - impact of clinical findings in late pregnancy. Man Ther. 2014 Jun;19(3):190-6. doi: 10.1016/j.math.2014.01.004. Epub 2014 Jan 22. PMID 24508067
- [Background] Malmqvist S, Kjaermann I, Andersen K, Okland I, Bronnick K, Larsen JP. Prevalence of low back and pelvic pain during pregnancy in a Norwegian population. J Manipulative Physiol Ther. 2012 May;35(4):272-8. doi: 10.1016/j.jmpt.2012.04.004. PMID 22632586
- [Background] O'Sullivan PB, Beales DJ. Diagnosis and classification of pelvic girdle pain disorders--Part 1: a mechanism based approach within a biopsychosocial framework. Man Ther. 2007 May;12(2):86-97. doi: 10.1016/j.math.2007.02.001. PMID 17449432
- [Background] Vermani E, Mittal R, Weeks A. Pelvic girdle pain and low back pain in pregnancy: a review. Pain Pract. 2010 Jan-Feb;10(1):60-71. doi: 10.1111/j.1533-2500.2009.00327.x. Epub 2010 Oct 26. PMID 19863747